CLINICAL TRIAL: NCT04335032
Title: A Randomised, Double-blind, Placebo Controlled Study of Eicosapentaenoic Acid (EPA-FFA) Gastro-resistant Capsules to Treat Hospitalised Subjects With Confirmed SARS-CoV-2
Brief Title: EPA-FFA to Treat Hospitalised Patients With COVID-19 (SARS-CoV-2)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPA-COV-001
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eicosapentaenoic acid gastro-resistant capsules (Experimental): Eicosapentaenoic acid free fatty acid (EPA-FFA) 500mg gastro-resistant capsules 2g daily (two capsules twice daily).
  One capsule of EPA-FFA gastro-resistant capsules contains 500mg EPA-FFA in a capsule containing gelatin, glycerol, sorbitol, titanium dioxide, FD&C blue No. 1, hypromellose phthalate, dibutyl sebacate.
  Interventions: Drug: Eicosapentaenoic acid gastro-resistant capsules
- Placebo (Placebo Comparator): Placebo capsules that cannot be visually differentiated from the active treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eicosapentaenoic acid gastro-resistant capsules — same as in arm/group description
  Other Names: Alfa
  Arms: Eicosapentaenoic acid gastro-resistant capsules
Drug: Placebo — same as in arm/group description
  Arms: Placebo

SUMMARY:
This is an double-blind, randomized, placebo controlled phase III study in hospitalized subjects with confirmed SARS-CoV-2.

DETAILED DESCRIPTION:
Recruitment SSubjects hospitalised or attended the hospital ED with a confirmed diagnosis of SARS-CoV-2, will be contacted.

Potential subjects will have the opportunity to ask any questions to the researchers.

A member of the research team will provide a copy of the information sheet to the subject, who will have the opportunity to ask any questions to the researchers.

Subjects expressing an interest in participating will be interviewed to explain the study in detail, and discuss the risks, benefits, goals and limitations of the study.

Screening Procedures. Potentially eligible subjects will provide informed consent prior to any study specific procedures being conducted.

Following the provision of informed consent, the subject's demographics and medical history especially that relating to SARS-CoV-2 will be documented.

A physical examination and checks on vital signs (BP, pulse, temperature, respiration) will be conducted. Female subjects of child-bearing potential will undergo a urine pregnancy test. A blood sample will be drawn for routine haematology and biochemistry. Subjects will undergo tests for oxygen saturation, PaO2/FiO2 and interleukin-6 (IL-6).

Subjects will be asked to provide details of any concomitant medications. Subjects with confirmed diagnosis of SARS-CoV-2, compliance with the inclusion and exclusion criteria and providing informed consent will be registered on the e-CRF to obtain a randomisation number.

Baseline/Randomisation A physical examination and checks on vital signs (BP, pulse, temperature, respiration) will be conducted. Subjects will undergo tests for oxygen saturation, PaO2/FiO2 and interleukin-6. Haematology and biochemistry test (from screening) results will be confirmed as being acceptable.

The study centre will dispense the IMP under blinded conditions according to a permuted block randomisation sequence (1:1 ratio for the two subject groups).

The subjects will be trained on the dosing and asked to administer two capsules twice daily for 4 weeks. Subjects will then be provided with IMP on a daily basis by a suitably qualified and delegated member of the Investigator's team, for the duration of the treatment phase.

Treatment Phase (Week 1-3) All subjects will receive standard of care treatment throughout the treatment phase on a day to day basis. This will include assessment of additional or alternative medication required for the treatment of SARS-CoV-2, requirement for intubation and invasive ventilation, requirement to transfer to intensive care unit or death.

On a weekly basis, a physical examination and checks on vital signs (BP, pulse, temperature, respiration) will be conducted. Subjects will undergo tests for oxygen saturation, PaO2/FiO2 and IL-6.

Subjects will be asked to provide details of any concomitant medications and changes in condition via adverse event (AE) query.

Week 4 A physical examination and checks on vital signs (BP, pulse, temperature, respiration) will be conducted. Subjects will undergo tests for oxygen saturation, PaO2/FiO2 and IL-6. Female subjects of child-bearing potential will undergo a urine pregnancy test. A blood sample will be drawn for routine haematology and biochemistry. Subjects will be asked to provide details of any concomitant medications and changes in condition via AE query.

Week 6 (Follow -up) 6 weeks after randomisation (or two weeks after early withdrawal), the subject will be contacted to check the occurrence of any other adverse events and review of medications. Haematology and biochemistry test (from week 4) results will be confirmed as being acceptable.

Adverse events will be assessed by spontaneous reports by subjects.

ELIGIBILITY:
Inclusion criteria:

The subject must satisfy the following criteria for entry into the study:

1. Male or female, aged 18 years and above.
2. Provide informed consent prior to any study specific procedure being conducted; for older patients who lack mental or physical capacity, next of kin or legal guardians will be allowed to provide consent on their behalf. This consent can be obtained remotely by telephone to the next of kin, or by a doctor with relevant experience in COVID-19 disease not directly involved in the study acting as the patient's advocate and then subsequently informing the next of kin (eg by a telephone call also offering them an opportunity to review and agree the ICF with them; the patient may then continue in the study or withdraw at a later date if the next of kin subsequently decides to withdraw consent).
3. Positive local approved test to confirm diagnosis of SARS-CoV-2 within 7 days prior to baseline.
4. Classified as moderate or severe based on the modified WHO/NIH baseline severity criteria. Moderate: evidence of lower respiratory disease by clinical assessment (e.g. signs or symptoms of lung infection) or by chest X-ray/CT/ultrasound imaging (e.g. viral pneumonia, lung infiltrates) and a saturation of oxygen (SaO2) ≥ 94% on room air at sea level. Severe: respiratory frequency >30 bpm, SaO2 < 94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) < 300 mmHg, or lung infiltrates >50%.
5. Hospitalised or attended the hospital ED due to clinical and/or virological diagnosis of SARS-CoV-2; subsequent follow up after screening may be carried out in hospital (hospitalised) or at a COVID-19 hospital OP clinic as clinically indicated at the investigator's discretion. Where it is not possible for the subject to attend a hospital OP clinic, then providing a suitably trained healthcare professional (eg part of the clinical research team) as directed by the investigator, is available to visit the subject at home to conduct the necessary clinical and SaO2 assessments and blood tests, subsequent assessments post-hospitalisation or ED visit may be conducted at the subject's home.

Exclusion criteria:

The subject will be excluded from the study if any of the following applies:

1. No symptoms or signs or lung imaging abnormalities of SARS-CoV-2.
2. On or clinically diagnosed as requiring intubation at screening.
3. On or clinically diagnosed as requiring mechanical ventilation at screening.
4. On or clinically diagnosed as requiring oxygen delivered by high flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5).
5. On or clinically diagnosed as requiring noninvasive positive pressure ventilation.
6. On or clinically diagnosed as requiring extracorporeal membrane oxygenation (ECMO).
7. Unable to swallow study capsules easily.
8. Known allergic reaction or intolerant to fish or fish oils.
9. Known allergic reaction to excipients of IMP.
10. Pregnant or breast-feeding at screening.
11. Taking other fish-oil supplements (e.g. cod liver oil) who are unwilling to stop them for the duration of the study.
12. Taking immunomodulators/immunosuppressants, including corticosteroids on entry into the study.
13. Used another investigational drug in the past 48 hours or 5 half-lives, whichever is longer, prior to Screening.
14. Participating in other clinical studies at the same time.
15. Evidence of multi-organ failure, SOFA score > 9.
16. Deemed, by the investigator, unlikely to be able to comply with the requirements of the protocol.
17. Deemed, by the investigator, likely to require transfer to the intensive care unit (ICU) or unlikely to survive for at least 48 hours.
18. Any gastro-intestinal symptoms at screening considered clinically significant.
19. Clinically significant abnormalities, which in the opinion of the investigator would significantly risk the safety of the subject or the main objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of EPA-FFA efficacy compared to placebo | 28 days
  Time to treatment failure during the 28-day treatment period. Treatment failure is defined as additional or alternative treatment required, or intubation and invasive ventilation, or transfer to intensive care unit, or death.

SECONDARY OUTCOMES:
Time to and amount of clinical improvement | 28 days
  To determine whether EPA-FFA gastro-resistant capsules decreases the time to and amount of clinical improvement as determined by the WHO 9-point ordinal scale during the study.
Change in recovery and survival rate | 28 days
  To determine whether EPA-FFA gastro-resistant capsules increases the number of subjects alive and discharged home without supplemental oxygen therapy.
Reduction of CRP and IL-6 | 28 days
  To determine whether EPA-FFA gastro-resistant capsules decreases CRP and IL-6 during the study.
Increase in IFN-γ | 28 days
  To determine whether EPA-FFA gastro-resistant capsules increases IFN-γ during the study
Reduction in proinflammatory chemokines and cytokines. | 28 days
  To determine whether EPA-FFA gastro-resistant capsules decreases other proinflammatory chemokines and cytokines.

OTHER OUTCOMES:
Safety - Vitals, AEs and Clinical lab parameters | throughout the study, about 3 months
  To evaluate the safety of EPA-FFA gastro-resistant capsules in the treatment of COVID-19 (SARS-CoV-2) by assessing subjects clinical lab parameters and vital signs, and the number and proportion of subjects with AEs.

CONTACTS AND LOCATIONS:
Locations (5):
- Hospital Universitario Vall d'Hebron, Barcelona, Spain
- United Kingdom (4):
  - Hull, Cottingham
  - UHCW, Coventry
  - NPH, Harrow
  - Rotherham NHS Foundation Trust, Rotherham

IPD SHARING:
Plan to Share IPD: No